CLINICAL TRIAL: NCT05101655
Title: Construction and Clinical Application of Microfluidic Exosome Chip for Early Diagnosis of Pulmonary Metastasis of Osteosarcoma
Brief Title: Construction of Microfluidic Exosome Chip for Diagnosis of Lung Metastasis of Osteosarcoma
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: (2020)LLS-NO395
Record Dates: First submitted 2021-10-07; First posted 2021-11-01 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Osteosarcoma; Pulmonary Metastases
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Use exosome microfluidic chips to establish a combination of exosome subgroup level (exosome barcode) markers for the early diagnosis of osteosarcoma lung recurrence, and establish the basis of microfluidic chip based exosome biomarker for monitoring the early therapeutic response of the second-line therapy for recurrent osteosarcoma.

DETAILED DESCRIPTION:
Osteosarcoma is the most common primary malignant bone tumor in adolescents, and lung metastasis is the main cause of its poor prognosis. Our previous data on the basis of second-line chemotherapy combined with VEGFRi targeted therapy for patients with lung metastases from osteosarcoma showed that some patients with early diagnosis of lung metastases may achieved long-term tumor-free survival upon prompt treatment. However, plasma biomarker for the early detection of recurrent osteosarcoma is still lacking to date. Our preliminary studies indicate that exosome is a potential source of liquid biomarker for the early diagnosis of osteosarcoma lung metastasis. We, therefore, have developed a microfluidic biochip based on nano-zinc oxide microcolumns. This chip can quickly and efficiently screen and capture exosomes and achieve quantitative and qualitative detection of exosome and its subgroups. This technology may be able to achieve early sensitive exosome quantification for lung metastasis of osteosarcoma. But the clinical efficacy and utility of the microfluidic chip based exosome detection for the early diagnosis osteosarcoma recurrence remains to be validated.

This research plan uses our newly developed microfluidic chip technology to capture and efficiently capture exosomes for quantitative and qualitative and marker screening, and establish a combination of exosome subgroups level as a biomarker for the early diagnosis of osteosarcoma lung metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy pathologically diagnosed as primary high-grade osteosarcoma (including ordinary osteosarcoma, vasodilatory osteosarcoma, small cell osteosarcoma, high-grade surface osteosarcoma);
2. Age no less than 12 years old and no older than 60 years old;
3. New-onset patients who have not received chemotherapy, radiotherapy, surgery, Chinese medicine and other treatments.
4. The primary site is the limbs and pelvis.

Exclusion Criteria:

1. Pathological diagnosis of surgical gross specimens except primary high-grade osteosarcoma;
2. Failure to collect circulating exosomes as planned;
3. Suffering from chronic diseases, which may lead to an increase in non-tumor-related circulating exosomes, such as autoimmune diseases , Chronic infections, etc.;
4. The use of targeted drugs may lead to a decrease in tumor-related circulating exosomes;
5. Withdrawal from the trial for any reason.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Surgical specimens and peripheral blood specimens of previous patients with osteosarcoma in the specimen bank,
  2. Patients who were diagnosed with osteosarcoma and were hospitalized in the Department of Orthopedics of Ruijin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
The association of disease recurrence with plasma levels of exosome and its subgroups. | through study completion, an average of 2 years
  After the patients were enrolled, MRI of the primary surgical site (enhanced if necessary), chest CT and bone scan were performed for the surveillance of disease recurrence according to the National Comprehensive Cancer Network (NCCN) guideline. The number of total plasma exosome as well as its subgroups (Vim, cluster of differentiation 44 (CD44), Integrins positive, etc.) were measured based on the microfluidic chip. The association of sarcoma recurrence with plasma exosome levels was then determined to validate the clinical efficacy of plasma exosome as a potential liquid biomarker.

SECONDARY OUTCOMES:
The change of plasma exosome level during the postoperative surveillance from baseline | through study completion, an average of 2 years
  The exosome and its subgroup levels were measured on the individual basis in comparison to the baseline to study the dynamic change of exosome during the postoperative surveillance from baseline.
The correlation of the therapeutic response with plasma levels of exosome and its subgroups. | at 1 month post-therapy
  For patients with recurrent disease who start second- or third- line therapy, the number of total plasma exosome as well as its subgroups (Vim, cluster of differentiation 44 (CD44), Integrins positive, etc.) were measured at 1 month post-therapy. We then assess the association of the exosome biomarker with the treatment response, as determined by Response Evaluation Criteria In Solid Tumours (RECIST) 1.1.
The correlation of microfluidic chip based exosome quantification with conventional approach | through study completion, an average of 2 years
  We investigate the correlation of microfluidic chip based plasma exosome levels with the conventional methodologies, such as Nanoparticle tracking analysis (NTA) and Western-blot

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China